CLINICAL TRIAL: NCT06258642
Title: Study of Irinotecan Liposome Combined With Anlotinib as Second-line Regimen in Patients With Small Cell Lung Cancer
Brief Title: Irinotecan Liposome Combined With Anlotinib as Second-line Regimen for SCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Doctor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-SCLC-K01
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Small Cell Lung Cancer Recurrent
Keywords: Small Cell Lung Cancer; liposomal irinotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — irinotecan sucrosofate; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan Liposome and anlotinib (Experimental): The treatment is continued until disease progression or intolerable toxicity
  Interventions: Drug: Irinotecan Liposome; Drug: Anlotinib

INTERVENTIONS:
Drug: Irinotecan Liposome — 70 mg/m^2 , d1, Q2W, iv
  Other Names: Irinotecan liposome injection
Drug: Anlotinib — 12 mg, qd, po for 2 consecutive weeks and then discontinued for 1 week.
  Other Names: Anlotinib hydrochloride

SUMMARY:
This study is a single arm, multi-center, prospective clinical trial. The purpose of this study is to evaluate the efficacy and safety of liposomal irinotecan combined with anlotinib hydrochloride for relapsed small-cell lung cancer, who have progressed on or less than 6 month after platinum-based first-line therapy.

DETAILED DESCRIPTION:
Patients will receive irinotecan liposome injection at 70 mg/m^2 intravenously, on Days 1 of every 14-day cycle and anlotinib (12 mg/day) for 2 consecutive weeks and then discontinued for 1 week. The treatment is continued until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged ≥18 and ≤75 years old;
* 2) Histologically or cytologically confirmed small cell lung cancer;
* 3) At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1;
* 4) Radiologically confirmed recurrence or progression within 6months after platinum-based, first-line chemotherapy or chemoradiation therapy;
* 5) Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
* 6) Expected survival of more than 3 months;
* 7) Recovered from the effects of any prior chemotherapy, surgery, radiotherapy or other anti-neoplastic therapy (recovered to no more than Grade 1 of CTCAE 5.0 criteria or baseline, with the exception of alopecia or other toxicity without safety concerns by the investigators' judgment);
* 8) Adequate major organ function, patients should meet the following criteria:

  ① Bone marrow function: absolute neutrophile count (ANC)≥1.5×109/L，platelet (PLT)≥100×109/L, hemoglobin (Hb)≥90g/L, white blood cell (WBC)≥3.0×109/L；

  ② Hepatic function: total bilirubin≤1.5×upper limit of normal value(ULN)；ALT and AST≤2.5×ULN，liver metastasis：≤5×ULN；

  ③ Renal function: serum creatinine ≤1.5×ULN and creatinine clearance rate ≥60 mL/min;

  ④ Coagulation function：Activated partial thromboplastin time(APTT)、International normalized ratio(INR)、prothrombin time (PT)≤1.5×ULN；

  ⑤ urine routines show urine protein < 2+(when urine protein >2+, urine protein quantity< 1.0 g during 24 hours before 7 days);
* 9) Patients fully understood and volunteered to participate in the study.

Exclusion Criteria:

* 1) Patients with large cell neuroendocrine lung carcinoma or combined small cell lung carcinoma;
* 2) Patients with asymptomatic central nervous system (CNS) metastases prior to enrollment or those who have CNS disease requiring increase in the dose of steroid. (Patients with controlled CNS metastasis can participate in the trial);
* 3) Patients with uncontrolled pleural effusion, abdominal effusion and pericardial effusion after repeated drainage or other treatment within 2 weeks prior to the first dose of this study, and those judged by the clinicians to be unsuitable for the study;
* 4) Diagnosed with any other cancer within the past 5 years (except for cured basal cell carcinoma and in situ cancer);
* 5) Patients who have received prior irinotecan/ liposomal irinotecan and anti-angiogenic drugs such as anlotinib and bevacizumab , etc.
* 6) Concomitant use of strong CYP3A4 inducers within 2 weeks or strong CYP3A4 inhibitors or strong UGT1A1 inhibitors within 1 week of the first dose of the study drug;
* 7) Patients who have received other anti-tumor treatments(including radiotherapy, chemotherapy, immunotherapy, etc.) within 4 weeks before the first dose;
* 8) Combined with uncontrolled systemic diseases, including unstable angina, myocardial infarction, congestive heart failure, severe ventricular arrhythmia , etc.
* 9) Severe pulmonary disease within 6 months prior to enrolment, such as interstitial pneumonia, pulmonary fibrosis, radiation induced pneumonitis requiring steroid therapy, and other moderate and severe lung diseases which affect lung function;
* 10) Arterial/venous thrombosis within 6 months prior to enrollment, e.g. cerebrovascular accident (include temporary ischemic attack), deep venous thrombosis, pulmonary embolism.
* 11) Symptoms or propensity to bleed within 3 months prior to screening (include gastrointestinal hemorrhage, ulcerative gastric bleeding, fecal occult blood 2+ or above, vasculitis);
* 12) Patients had undergone major surgical procedure(except for diagnostic surgery) within 4 weeks before dosing or was scheduled to receive major procedure during the study;
* 13) unhealed wounds, ulcers or fractures;
* 14) Imaging showed tumors have involved important blood vessels or by investigators determine likely during the follow-up study and cause fatal hemorrhage;
* 15) Active and uncontrolled bacterial, viral, fungal infection requiring systemic treatment;
* 16) Active hepatitis B/C, or HIV infection;
* 17) Known intolerance or allergy to therapeutic drugs and their excipients;
* 18) Clinically significant gastrointestinal disorder, including hepatic disorders, bleeding, inflammation, occlusion, or diarrhea > grade 1;
* 19) Pregnant or breast feeding;
* 20) Patient is not suitable for the study in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | From date of first dose until the date of first documented progression, assessed up to 24 months
  To evaluate anti-tumor efficacy

SECONDARY OUTCOMES:
Disease control rate (DCR) | From date of first dose until the date of first documented progression, assessed up to 24 months
  To evaluate anti-tumor efficacy
Duration of Response(DoR) | From date of first dose until the date of first documented progression, assessed up to 24 months
  To evaluate anti-tumor efficacy
Progression-Free Survival (PFS) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To evaluate anti-tumor efficacy
Overall Survival (OS) | From date of first dose until the date of death from any cause , assessed up to 24 months
  To evaluate anti-tumor efficacy
Incidence and severity of adverse events | date of the first dose to 28 days after permanent treatment termination
  To evaluate the safety

CONTACTS AND LOCATIONS:
Overall Officials: Jialei Wang, Doctor, Principal Investigator — Fudan University
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No